CLINICAL TRIAL: NCT05292989
Title: A Personalised Approach Utilising the Frailty Index to Empower Consumers to Make Informed Decisions About Having a Colonoscopy to Avoid Low Value Care. A Prospective Randomized Controlled Trial.
Brief Title: A Personalised Approach Utilising the Frailty Index to Empower Consumers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Alexandra Hospital, Brisbane, Australia (Other)
Responsible Party: Principal Investigator, Gerald Holtmann, Director of Gastroenterology & Hepatology, Princess Alexandra Hospital, Brisbane, Australia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Frailty Study
Record Dates: First submitted 2022-03-01; First posted 2022-03-23 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Gastrointestinal Diseases
Keywords: colonoscopy surveillance
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial design
Who Masked: Outcomes Assessor
Masking Description: Deidentified data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1- Personalised tailored approach (Experimental): If patients are assigned to this group they will be asked to complete a frailty assessment which includes the Fraility Index short form, an assessment of grip strength, time to complete 5 sit-to-stands, balance test, and gait speed along with some questionnaires on comorbid medical condition. The treating Gastroenterologist will then go through the results of the frailty assessment with the patient and based on this information will discuss the benefits and risks associated with having a surveillance colonoscopy. The patient will then decide if they would like to go ahead with a surveillance colonoscopy and the treating Gastroenterologist will provide further advice as required. The frailty assessment is intended to be done at the time of the appointment with the specialist. However, operational requirements may dictate that e.g. a telehealth delivered occasion of service is done at a separate date.
  Interventions: Other: Frailty Assessment
- Group 2- Standard Care (Placebo Comparator): Patients assigned to this group will discuss the benefits and risks associated with having a surveillance colonoscopy with the treating Gastroenterologist and will decide whether to proceed with the colonoscopy.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Frailty Assessment — Personalised (tailored) approach that includes assessment of frailty and structured information provided to the consumer
  Arms: Group 1- Personalised tailored approach
Other: Standard Care — Standard care practice
  Arms: Group 2- Standard Care

SUMMARY:
Frailty is a common clinical syndrome in older adults that may carry an increased risk for poor health outcomes including falls, hospitalisation, and mortality. Having a colonoscopy can be associated with potential adverse outcomes in frail patients. At present, however, frailty is not routinely assessed in gastroenterological clinical practice. In a prospective randomised controlled study consenting patients over 65 years at the Princess Alexandra Hospital will receive either a) personalised (tailored) approach that includes assessment of frailty and structured information provided to the consumer or b) current standard practice in regards to having a surveillance colonoscopy to determine the effects on patient satisfaction and percentage of colonoscopies avoided.

DETAILED DESCRIPTION:
Frailty is a common clinical syndrome in older adults that may carry an increased risk for poor health outcomes including falls, hospitalisation, and mortality. Having a colonoscopy can be associated with potential adverse outcomes in frail patients. At present, however, frailty is not routinely assessed in gastroenterological clinical practice. In a prospective randomised controlled study consenting patients over 65 years at the Princess Alexandra Hospital will receive either a) personalised (tailored) approach that includes assessment of frailty and structured information provided to the consumer or b) current standard practice in regards to having a surveillance colonoscopy to determine the effects on patient satisfaction and percentage of colonoscopies avoided. It is expected that engagement with patients and clinicians in regards to frailty will address expectations and subsequently support the ability of patients/consumers and clinicians to make informed decisions that minimise risks and maximise benefits in regards to surveillance colonoscopies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 65 years of age
* Ability to understand the study instructions and answering questionnaires

Exclusion Criteria:

* Inability to consent or participate in the assessments (e.g. frailty assessment) that are required as part of this project.
* Lack of informed consent

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-14 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with the respective outpatient service. | Week 0
  'Based only upon your recent experience when you received a consultation in relation to a potential future endoscopic test, how likely are you to recommend the respective health care organization (PAH or RWBH) to a friend, family member or colleague?.'
  Please rate your experience on a scale of 1 to 10, where 1 is extremely unlikely and 10 extremely likely.
Patient satisfaction questions | Week 0
  Patients will be asked
  Overall, how would you rate the care you received? 1. Very good 2. Good 3. Adequate 4. Poor 5. Very poor
  Were you involved as much as you wanted to be in decisions about your care and treatment? 1. Yes, definitely 2. Yes, to some extent 3. No, not enough
  How much information about your condition or treatment was given to you? 1. The right amount 2. Too much 3. Not enough
Comprehensive Endoscopy Satisfaction Tool | Week 2-4 After colonoscopy procedure
  This captures the overall satisfaction with the service events (endoscopic procedure and relevant components including the pre-procedure assessment). Higher scores greater satisfaction
Percentage of consumers in the intervention and control group that are referred for a surveillance colonoscopies who decide not have the procedure based upon the information provided. | Week 0-2 after consultation with doctor
  • Percentage of consumers in the intervention and control group that are referred for a surveillance colonoscopies who decide not have the procedure based upon the information provided.

SECONDARY OUTCOMES:
Number of participants with colorectal cancer related morbidity | Colorectal cancer related morbidity within 5 years of the referral
  The number of participants with colorectal cancer related morbidity within 5 years of the referral- including number of patients with clinical diagnoses, hospitalizations, emergency presentations, surgeries, medications
Number of participants with non colorectal cancer related mortality information within 5 years of the referral | Non colorectal cancer related mortality information within 5 years of the referral
  The number of participants with non colorectal cancer related mortality information within 5 years of the referral - including number of patients with clinical diagnoses, hospitalizations, outpatient visits, emergency presentations, surgeries

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Alexandra Hospital, Woolloongabba, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No